CLINICAL TRIAL: NCT03898297
Title: Imaging mGluR5 and Synaptic Density in Psychiatric Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000020186; 1R01MH116657-01A1 (NIH); 1K23DA045957-01 (NIH)
Record Dates: First submitted 2018-12-21; First posted 2019-04-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Healthy
Keywords: Depression; Bipolar; Mood disorder; PET; mGluR5; glutamate system; MRI
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression; Mood Disorders | interventions — 1-((3-(methylpyridin-4-yl)methyl)-4-(3,4,5-trifluorophenyl)pyrrolidin-2-one

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control: 60 psychiatrically-healthy subjects will be enrolled as controls may participate in MRI or fMRI, [1H]MRS and/or [13C]MRS, [18F]FPEB and/or [11C]APP311 PET scans, cognitive testing
  Interventions: Radiation: [18F]FPEB; Radiation: [11C]APP311
- MDD: 30 subjects with major depressive disorder (MDD) may participate in MRI or fMRI, [1H]MRS and/or [13C]MRS, [18F]FPEB and/or [11C]APP311 PET scans, cognitive testing
  Interventions: Radiation: [18F]FPEB; Radiation: [11C]APP311
- Bipolar: 30 subjects with bipolar disorder may participate in MRI or fMRI, [1H]MRS and/or [13C]MRS, [18F]FPEB and/or [11C]APP311 PET scans, cognitive testing
  Interventions: Radiation: [18F]FPEB; Radiation: [11C]APP311

INTERVENTIONS:
Radiation: [18F]FPEB — Radiotracer: [18F]FPEB
Radiation: [11C]APP311 — Radiotracer: [11C]APP311, [11C]UCB-J
  Other Names: [11C]UCB-J

SUMMARY:
This research study is designed to look at the involvement of the glutamate system and synaptic density in depression and bipolar disorder. Each participant will undergo a screening appointment to determine study eligibility. Thereafter, the study will take 2 or 3 visits depending on schedule availability and will consist of a combination of one magnetic resonance imaging (MRI) or functional magnetic resonance imaging (fMRI) scan, one proton magnetic resonance spectroscopy (MRS) and/or one C13 MRS scans, and up to two positron emission tomography (PET) scans. Participants will also participate in cognitive testing. Depending on camera time, staff availability and subject schedule, total study participation may last 1-2 months.

DETAILED DESCRIPTION:
With the recent advancements in the positron emission tomography (PET) and radioligand development, the investigators are now able to image and quantify the metabotropic glutamatergic system (mGluR5) in vivo in human subjects. The investigators propose a novel investigation using [18F]FPEB in depression and bipolar disorder to obtain critical data to advance the understanding of the etiology of depression and bipolar disorder and its associated symptoms of cognitive dysfunction. The findings with mGluR5 by themselves are limited. Changes in mGluR5 availability could be due to changes in synaptic density. Recently, the Yale PET center synthesized a new radioligand [11C]UCB-J (referred to as [11C]APP311 at the Yale University PET Center) that binds to synaptic vesicle glycoproteins (SV2A), which represent the number of synapses in the brain. Thus, the investigators will also measure synaptic density in the brain and relate to mGluR5 availability.

Aim 1: To determine mGluR5 availability with mood disorders compared to healthy controls as measured with PET brain imaging using [18F]FPEB.

Hypothesis 1: decrease in mGluR5 availability in individuals with mood disorders in regions responsible for emotional and cognitive processes, including the amygdala, hippocampus, thalamus, anterior cingulate, and frontal cortices.

Aim 2: To determine if glutamate cycling in individuals with mood disorders is altered as compared to healthy controls as measured with [1H]MRS and [13C]MRS.

Hypothesis 2: increase in glutamate number in individuals with mood disorders as compared to controls.

Aim 3: To determine if the PET alterations in the glutamatergic system of depressed individuals are associated with cognitive deficits observed in depression, including concentration, attention, and memory (cognitive testing performance), and distractibility and startle.

Hypothesis 3: positive relationship between mGluR5 availability and cognitive functioning, such that individuals with higher receptor availability will perform better on tests of concentration, attention, memory, distractibility, and startle than individuals with lower receptor availability.

Aim 4: To examine whether changes in mGluR5 availability are dependent on state, or whether the lower availability is due to trait.

Hypothesis: normalization (or increase) in mGluR5 availability in euthymia as compared to depressed state.

Aim 5: To examine synaptic density changes associated with mood disorders using [11C]APP311 Hypothesis 5: lower synaptic density in individuals with MDD and bipolar disorder (BD), and associations between synaptic density changes and mood severity. Investigators also hypothesize there might be a relationship between synaptic density and mGluR5 availability.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

18-80 years old English speaking

-Inclusion criteria for healthy controls: no current, or history of any DSM-5 diagnosis

* Inclusion criteria for MDD subjects clinical diagnosis of major depressive disorder
* Inclusion criteria for bipolar subjects clinical diagnosis of bipolar disorder

Exclusion Criteria:

* Current or past significant medical, neurological, or metabolic disorder
* history of head injury that led to significant long term decline in cognitive abilities as seen by decline in grades or work performance
* history of significant medical illness such that would contraindicate study participation based on above criteria and PI/MD history review
* Active, significant suicidal ideation
* Implanted metallic devices or any MR contraindications
* women who are pregnant or breastfeeding
* Met Diagnostic and Statistical Manual of Mental Disorders(DSM)-5 criteria for mild substance use disorder in the past 6 months or moderate to severe substance use disorder within the past year (except marijuana or nicotine)
* history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year
* Current, past, or anticipated exposure to radiation in the work place within one year of proposed research PET scans
* Blood donation within 8 weeks of the start of the study
* History of a bleeding disorder or currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 60 psychiatrically-healthy controls 30 MDD 30 bipolar
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-01-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
mGluR5 availability using [18F]FPEB | Through study completion date: 5 years
  Glutamate (major excitatory neurotransmitter)is widespread throughout the brain & likely modulates some symptoms present in individuals w/mood disorders. Glutamate neurotransmission is regulated by ionotropic & the G-protein coupled metabotropic glutamate receptors (mGluR) which are divided into 3 groups: group I (mGluR1 and 5), group II (mGluR2 and 3) & group III (mGluR4, 6, 8). The group I mGluRs couple to phospholipase C, & stimulate cyclic AMP formation & arachidonic acid release & thus impact neuroplasticity, neuronal excitability, synaptic transmission & gene expression. mGluR5 receptors are located post synaptically & on glia,& have highest density in hippocampus, intermediate in caudate/putamen, cerebral cortex, deep cerebellar nuclei, & thalamus, & lowest in the cerebellum. mGluR5 are considered to be pivotal in the functioning of the glutamatergic system especially as it pertains to cognitive performance.
  [18F]FPEB: high affinity radiotracer used to image mGluR5 receptor.
Synaptic density using [11C]APP311 | Through study completion date: 5 years
  Synaptic density differences using [11C]APP311 between individuals with mood disorders compared to healthy controls.
  Synaptic density and [11C]APP311: There is strong preclinical evidence showing that chronic stress and depression lead to structural changes, which include neuronal atrophy, reduced synaptic density and cell loss. [11C]APP311 (also referred to as [11C]UCB-J) was developed at the Yale University PET Center as a novel PET radioligand for synaptic vesicle glycoprotein 2A (SV2A). SV2A is an integral membrane protein located in presynaptic vesicle membranes, similar to synaptophysin (SYN). SV2 has 3 isoforms, with SV2A being the only isoform which is ubiquitously located in synaptic vesicles across the brain. Thus, PET quantification of SV2A signal may be an excellent in vivo biomarker of synaptic density.

SECONDARY OUTCOMES:
glutamate cycling using MRS | Through study completion date: 5 years
  alterations in glutamate cycling in individuals with mood disorders compared to healthy controls using [1H]MRS and [13C]MRS
  [1H]MRS: proton Magnetic Resonance Spectroscopy (MRS) [13C]MRS: baseline spectra obtained then [13C]glucose administered at a rate to raise the fractional 13C enrichment of the plasma glucose quickly to 60% and maintain it constant for 120 minutes, with a plasma glucose concentration between 150 and 200 mg/dl. The 13C MRS measurements will continue throughout the infusion of glucose. These data will be analyzed using a metabolic model to derive the rates of oxidative glucose metabolism and glutamate neurotransmitter cycling.
Cognitive Functioning Assessed with CogState Software | Through study completion date: 5 years
  relationship between cognitive functioning and mGluR5 availability in individuals with mood disorders compared to healthy controls.
  Cognitive functioning: the way people think, remember, and process information. Utilizing CogState software.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Esterlis, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University PET Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No